CLINICAL TRIAL: NCT03873233
Title: Flow Controlled Ventilation With the Evone Ventilator and Tritube Versus Volume Controlled Ventilation: A Clinical Pilot Study Describing Oxygenation, Ventilation and Haemodynamic Variables
Brief Title: Flow Controlled Ventilation (FCV) With the Evone Ventilator and Tritube Versus Volume Controlled Ventilation (VCV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Joke De Wachter, data manager, University Hospital, Antwerp
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18/45/512
Record Dates: First submitted 2019-02-07; First posted 2019-03-13 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Ventilation

STUDY DESIGN:
Intervention Model Description: Patients undergoing craniotomy will be ventilated during surgery using both conventional VCV and FVC modes. Standard baseline VCV is used for induction and stabilization of anesthesia. The order of ventilation mode is randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Volume Controlled Ventilation (Active Comparator): Volume Controlled Ventilation with Aisys Carestation ventilator and normal endotracheal tube'
  Interventions: Device: Aisys Carestation ventilator and normal endotracheal tube
- Flow Controlled Ventilation (Active Comparator): Flow Controlled Ventilation with Evone ventilator and Tritube
  Interventions: Device: Evone ventilator and Tritube

INTERVENTIONS:
Device: Aisys Carestation ventilator and normal endotracheal tube — Fraction of Inspired Oxygen (FIO2) 0.3 End Expiratory Pressure (EEP) at +5 cm H2O Ratio of duration of inspiration to the duration of expiration (I:E ratio) 1:1 Tidal Volume: 6 mL/kg Zero inspiratory pause Respiratory frequency will be adapted to produce an End-Tidal CO2 35-40 mmHg
  Arms: Volume Controlled Ventilation
Device: Evone ventilator and Tritube — Fraction of Inspired Oxygen (FIO2) 0.3 Ratio of duration of inspiration to the duration of expiration (I:E ratio) 1:1 End Expiratory Pressure (EEP) at +5 cm H2O Flow: start with 10 L/min and adjusted along with the peak inspiratory pressure to produce a tidal volume of 6 mL/kg and End-Tidal CO2 35-40 mmHg
  Arms: Flow Controlled Ventilation

SUMMARY:
The Evone® ventilator is a new device capable of lung ventilation through a narrow-bore cannula, the Tritube.Two ventilation modes are possible: high frequency jet ventilation (HFJV) and flow-controlled ventilation (FCV). In this prospective pilot study the efficacy of FCV using the Evone® ventilator and Tritube is investigated when compared with Volume Controlled Ventilation (VCV) via a normal tracheal tube.

DETAILED DESCRIPTION:
The Evone® (Ventinova Medical, Eindhoven, The Netherlands) is an automated mechanical ventilator providing pulmonary ventilation by generating a continuous flow into the patient's lungs during inspiration as well as a continuous flow during expiration (flow controlled ventilation, FVC). FCV is a relatively new concept in which ventilation via the Tritube (Ventinova), an ultrathin endotracheal tube, has been made possible due to active suctioning of gas from the lungs during expiration (expiratory ventilation assistance, (EVA)). Adjustable parameters that govern the FCV cycle are: Inspiration Flow, Inspiratory:Expiratory ratio (I:E ratio), maximum tracheal pressure (PMAX) and end expiratory pressure (EEP). Measured parameters are: end-tidal carbon dioxide partial pressure (PE'CO2 ) as measured by capnography, Minute Volume, Peak Tracheal Pressure, End Expiratory Pressure, Respiratory Frequency, I:E ratio and Tidal Volume ( VT). The ventilator screen continuously displays a capnograph with end-tidal CO2, intra-tracheal pressure and inspiratory tidal volume waveforms. In FCV mode, inspiration occurs with the pre-set, constant inspiratory flow until the intratracheal pressure reaches the pre-set value. Assisted expiration then occurs until the pre-set EEP is reached. Expiratory flow is controlled in such a way to achieve a mainly linear reduction in tracheal pressure, whilst ensuring the set I:E ratio. There are no inspiratory or expiratory pauses and EVA does not result in negative tracheal pressures. Thus, minute volume is determined by the set flow rate and the I:E ratio. The set inspiratory peak and end expiratory pressures determine the tidal volumes. Ventilatory frequency is a result of these parameter settings.

The Tritube is a 40 centimeter long narrow diameter cuffed tracheal tube (internal diameter 2.4 millimeter, outer diameter 4,4 millimeter) that can be used with either the manual Ventrain® or automated Evone® ventilator. It consists of three lumens: a ventilatory channel with Murphy eye, a channel for airway pressure measurement and a channel for inflating the high volume, low pressure polyurethane cuff. Preliminary data suggests that Evone® not only provides adequate ventilation via the Tritube, but in comparison with conventional modes of ventilation (volume-controlled, pressure-controlled modes) may result in improved alveolar gas distribution, ventilation/perfusion matching, respiratory mechanics and oxygenation. In this prospective pilot study the efficacy of FCV using the Evone® ventilator and Tritube is investigated when compared with VCV (Aisys Carestation, GE Healthcare, WI, USA) via a normal tracheal tube.

All participants meeting inclusion criteria and having signed Informed Consent will undergo anesthesia and monitoring as per standard of care for the designated surgical procedure (5 lead ECG, non-invasive blood pressure cuff, saturation monitor). Neuromuscular blockade will be monitored by use of the TOF Watch®SX (train-of- four). Depth of anesthesia will be monitored by use of NeuroSENSE ®NS 701 Monitor( NeuroWave Systems incorporated - Cleveland Heights,OH). Following placement of a peripheral intravenous infusion, induction of standard intravenous anesthesia (propofol/remifentanil) and deep neuromuscular relaxation (rocuronium) will be established. Following 3 minutes of preoxygenation (Fractional end-tidal oxygen concentration (FE'O2> 0.9), patients will be intubated with a conventional cuffed tracheal tube cut to 24 centimeter length via oral route and ventilated in standard VCV mode with Fractional Inspired Oxygen concentration (FIO2) at 0.3 percent, Positive End Expiratory Pressure (PEEP + 5cmH2O) and frequency (f) of 12 breaths per minute. Tidal volume will be adjusted to ensure normocapnia. A radial arterial catheter will be placed and attached to a FloTrac sensor and Vigileo monitor ( Edwards Lifesciences, Irvine CA, USA) for continuous measuring of arterial blood pressure and cardiac output. It will facilitate blood gas sampling. Bladder temperature is monitored by means of a urinary catheter and patient is kept warm by means of a warming mattress and air warming blanket. After this preparation phase and prior to start of surgery, each subject will undergo two randomly allocated study periods: one with VCV, the other with FCV. In both cases FIO2 will be 0.3%, EEP at +5 cmH2O and I:E 1:1. Before starting the study protocol all subjects will be pre-oxygenated with 100% Oxygen for three minutes and undergo a recruitment manoeuvre. The recruitment manoevre will be conducted as follows: respiratory rate 12 breaths/minute, tidal volume 6mL/kg, initial PEEP 5cm H2O, with PEEP increasing in 5cm H2O increments to 15cm H2O per 5 breaths and then in decremental steps of 5cm H2O per 5 breaths back to 5 cm H2O PEEP. Peak pressure will be limited to 35 cm H2O.The respiratory circuit will then be disconnected for one minute. This provides sufficient time for placement of the Tritube through the tracheal tube when the subject is randomised to FCV in the first study period. For subjects initially randomised to VCV, VCV will be continued after this sham manoevre. Data collection starts after 15 minutes to allow stabilisation of respiratory and hemodynamic variables. Following data collection, a second 3 minutes pre-oxygenation period with recruitment manoevre and 1 minute apnea will be used before switching to the second ventilation mode.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for craniotomy in the supine position due to intracranial neoplasia
* American Society of Anesthesiologists (ASA) Class ≤ 3
* BMI < 30

Exclusion Criteria:

* Respiratory disease
* Severe cardiovascular disease
* Non-sinus rhythm
* Poorly controlled hypertension
* Patients with known allergies for rocuronium, propofol or remifentanil
* Emergency procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Observation of systemic arterial oxygen partial pressure (PaO2) values in both ventilation modes during normocapnia (PE'CO2 35-40 mm Hg) . | Following stable ventilation for 15 minutes in randomised ventilation modus, data collection starts and ends before start of surgery.
  Following stable ventilation for 15 minutes with respect to randomised ventilation mode, arterial blood gas will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium